CLINICAL TRIAL: NCT07276100
Title: Fecal Microbiota Transplantation to RESCUE Patients With Unresectable Hcc Progressors to First Line Therapy With AtezolizUmaB and Bevacizumab
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Fabio Piscaglia, Head of Division of Internal Medicine, Hepatobiliary and Immunoallergic Diseases, IRCCS Azienda Ospedaliero-Universitaria di Bologna , Clinical Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RESCUE-HUB; 2023-510504-45-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-25; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hepato Cellular Carcinoma (HCC)
Keywords: hepato cellular carcinoma; atezolizumab; microbiota; fecal microbiota trasplant
MeSH Terms: interventions — Fecal Microbiota Transplantation; atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental (Experimental): Fecal microbiota transplantation (FMT) + atezolizumab (1200 mg flat dose) and bevacizumab (15 mg/kg) Q3W
  Interventions: Other: Fecal microbiota transplantation (FMT); Drug: Atezolizumab & Bevacizumab

INTERVENTIONS:
Other: Fecal microbiota transplantation (FMT) — Fecal microbiota transplantation (FMT)
Drug: Atezolizumab & Bevacizumab — Atezolizumab & Bevacizumab

SUMMARY:
The purpose of this study is to evaluate whether fecal microbiota transplantation (FMT), when administered in combination with atezolizumab and bevacizumab, can improve treatment response in participants with hepatocellular carcinoma (HCC) whose disease has progressed during prior atezolizumab-bevacizumab therapy. The study will also assess the safety and feasibility of this treatment strategy.

Primary Objective:

To determine whether FMT can restore or enhance response to atezolizumab and bevacizumab following disease progression.

Participants will:

Receive a fecal microbiota transplantation (FMT).

Resume treatment with atezolizumab and bevacizumab, administered every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form.
2. Age ≥ 18 years.
3. Tolerance to first-line treatment for HCC with atezolizumab plus bevacizumab, defined as absence of adverse events requiring permanent discontinuation of either drug.
4. Ability to comply with all study procedures, in the investigator's judgment.
5. Unresectable hepatocellular carcinoma with early disease progression on first-line atezolizumab + bevacizumab (within 4 months of treatment initiation).
6. At least one untreated measurable lesion per RECIST 1.1.
7. ECOG Performance Status 0-1.
8. Child-Pugh class A.
9. Adequate hematologic and end-organ function (laboratory values obtained within 7 days prior to enrollment), defined as follows:

   1. ANC ≥ 1.5 × 10⁹/L (1500/µL), without G-CSF support.
   2. Lymphocyte count ≥ 0.5 × 10⁹/L (500/µL).
   3. Platelet count ≥ 60 × 10⁹/L (60,000/µL), without transfusion.
   4. Hemoglobin ≥ 90 g/L (9 g/dL); transfusion allowed if last transfusion ≥ 3 weeks prior.
   5. AST, ALT, and ALP ≤ 5 × ULN.
   6. Total bilirubin ≤ 3 × ULN.
   7. Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min (Cockcroft-Gault).
   8. Serum albumin ≥ 28 g/L (2.8 g/dL), without infusion supplementation in previous 2 months.
   9. INR and aPTT ≤ 1.5 × ULN.
10. Women of childbearing potential:

    a. Agree to remain abstinent or use effective contraception (failure rate <1%/year) during treatment and for 5 months after last atezolizumab dose and 6 months after last bevacizumab dose.

    b. Agree to refrain from donating eggs during this period.
11. Men with female partners of childbearing potential:

    1. Agree to remain abstinent or use a condom plus an additional contraceptive method (combined failure rate <1%/year) during treatment and for 6 months after last bevacizumab dose.
    2. Agree to refrain from donating sperm during this period.

Exclusion Criteria:

1. History of leptomeningeal disease or brain metastases.

2. Active or prior autoimmune disease or immune deficiency (e.g., myasthenia gravis, myositis, autoimmune hepatitis, SLE, RA, IBD, antiphospholipid syndrome, Wegener, Sjögren, Guillain-Barré, MS), except:

1. Autoimmune hypothyroidism on replacement therapy.
2. Controlled Type 1 diabetes on insulin.
3. Dermatologic-only autoimmune diseases (eczema, psoriasis, lichen simplex chronicus, vitiligo) if:

   1. Rash <10% BSA. 2. Well-controlled on low-potency topical steroids. 3. No exacerbations requiring systemic therapy within 12 months.

   3. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on CT (radiation pneumonitis in field allowed).

   4. Active tuberculosis.

   5. Significant cardiovascular disease within 3 months (NYHA ≥ II, MI, CVA), unstable arrhythmia, or unstable angina.

   6. Congenital long-QT syndrome or QTcF >500 ms at screening.

   7. Active advanced malignancy other than HCC within 1 year.

   8. Prior severe adverse reaction to atezolizumab or bevacizumab unmanageable with low-dose steroids or requiring discontinuation.

   9. Uncorrectable electrolyte abnormalities (K, Ca, Mg).

   10. Major surgery within 4 weeks or planned major surgery during study.

   11. Severe infection within 4 weeks (including hospitalization, bacteremia, severe pneumonia).

   12. Therapeutic oral/IV antibiotics within 2 weeks (prophylactic antibiotics allowed). All within 30 days has to be recorded in eCRF.

   13. Prior allogeneic stem cell or solid organ transplantation.

   14. Any condition or laboratory abnormality posing excessive risk or interfering with study results.

   15. Live attenuated vaccine within 4 weeks before treatment or planned during or 5 months after atezolizumab.

   16. Severe allergic or anaphylactic reaction to humanized antibodies or fusion proteins.

   17. Hypersensitivity to CHO cell products or components of atezolizumab or bevacizumab.

   18. Pregnancy or breastfeeding; intent to become pregnant during treatment or post-treatment windows.

Pregnancy test required within 14 days pre-treatment.

19. Fibrolamellar HCC, sarcomatoid HCC, or combined HCC-cholangiocarcinoma.

20. Untreated or high-risk esophageal/gastric varices. EGD required; prophylactic treatment mandated.

21. Variceal bleeding within 6 months.

22. Clinically evident ascites.

23. Episode of encephalopathy within 3 months.

24. HBV/HCV co-infection.

25. Patients with prior HCV but negative HCV RNA are considered non-infected.

26. Prior systemic therapy for advanced HCC other than first-line atezolizumab + bevacizumab.

27. Systemic immunostimulatory agents (e.g., interferon, IL-2) within 4 weeks or 5 half-lives.

28. Symptomatic, untreated, or actively progressing CNS metastases. Eligible only if all criteria are met: extracranial measurable disease, no hemorrhage history, lesions limited to cerebellum/supratentorial region, no progression post-therapy, no recent RT/surgery, no steroid requirement, stable anticonvulsants, new lesions treated before enrollment.

29. Uncontrolled tumor-related pain; symptomatic lesions requiring RT must be treated first.

30. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring ≥ monthly drainage.

Indwelling catheters allowed.

31. Uncontrolled or symptomatic hypercalcemia.

32. Investigational therapy (other than atezolizumab + bevacizumab) within 28 days.

33. Systemic immunosuppressive therapy within 2 weeks, except:

1. Acute, low-dose, or one-time pulse steroids.
2. Mineralocorticoids, inhaled steroids, low-dose steroids for adrenal insufficiency/orthostatic hypotension.

   34. Uncontrolled hypertension (SBP >150 mmHg and/or DBP >100 mmHg on multiple readings).

   35. Prior hypertensive crisis or hypertensive encephalopathy.

   36. Significant vascular disease within 6 months.

   37. Hemoptysis >2.5 mL within 1 month.

   38. Bleeding diathesis or significant coagulopathy.

   39. Current or recent (within 10 days of first dose of study treatment) use of aspirin >325 mg/day or treatment with dipyramidole, ticlopidine, clopidogrel, and cilostazol.

   40. Current or recent (within 10 days prior to study treatment start) use of full dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic (as opposed to prophylactic) purpose. Prophylactic anticoagulation for the patency of venous access devices is allowed provided the activity of the agent results in an INR < 1.5 x ULN and aPTT is within normal limits (ratio <1.5) within 14 days prior to initiation of study treatment.

   41. Core biopsy or minor surgery (except vascular access) within 3 days of first bevacizumab dose.

   42. History of abdominal or tracheoesophageal fistula, GI perforation, or intra-abdominal abscess within 6 months.

   43. History of intestinal obstruction and/or clinical signs or symptoms of GI obstruction including subocclusive disease related to the underlying disease or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding prior to initiation of study treatment. Patients with signs/symptoms of sub-/occlusive syndrome/intestinal obstruction at time of initial diagnosis may be enrolled if they had received definitive (surgical) treatment for symptom resolution.

   44. Abdominal free air not explained by procedure or surgery.

   45. Serious non-healing wound, ulcer, or untreated bone fracture.

   46. Metastatic disease involving major airways/blood vessels or large mediastinal masses (<30 mm from carina).

   Portal/hepatic vein invasion allowed.

   47. Intra-abdominal inflammatory process (e.g., complicated PUD, diverticulitis, colitis) within 6 months.

   48. Radiotherapy within 28 days (or abdominal/pelvic RT within 60 days), except palliative bone RT within 7 days.

   49. Local liver therapy (RFA, ethanol, cryoablation, HIFU, TACE, TAE, SIRT) within 28 days or incomplete recovery.

   50. Major surgery, open biopsy, abdominal surgery, abdominal intervention, or significant trauma within the specified windows or unresolved from such events.

   51. Chronic daily NSAID use, except aspirin <325 mg/day. Occasional use allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
incidence of adverse events of grade > 3 | through study completion, approximately 3 years
disease control rate | 12 weeks after FMT

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS AOU di Bologna Policlinico di Sant'Orsola, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No